CLINICAL TRIAL: NCT05382546
Title: A Phase 1, Open-label Pharmacokinetic Study of Intravenous NTM-001 (A Novel Formulation of Ketorolac Tromethamine Applied by Continuous Intravenous Infusion From A Pre-Mixed Bag) in Healthy Chinese Subjects
Brief Title: A Pharmacokinetic Study of Intravenous NTM-001 in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nuance Pharma (shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTM-001-AHC001
Record Dates: First submitted 2022-05-10; First posted 2022-05-19 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ketorolac Tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- NTM-001 Treatment Arm (Experimental): NTM-001 loading dose of 12.5 mg administered over approximately 60 seconds, followed by a continuous IV infusion at a rate of 3.5 mg/h for 24h, by a pre-programmed infusion pump.
  Interventions: Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Ketorolac Tromethamine — Ketorolac tromethamine, alcohol free formulation, 1.0 mg/mL in saline solution (~0.9% NaCl) adjusted to a pH of ~7.4. Contained in a sterile, polyolefin bag filled with 125 mL of NTM-001.
  Other Names: NTM-001 (Ketorolac Tromethamine IV Continuous Infusion)

SUMMARY:
This will be a single center, open-label phase 1 study in healthy Chinese subjects. A total of up to 16 subjects may be enrolled to achieve a total target of 12 evaluable subjects. A full dose for NTM-001 will be defined as a 12.5 mg IV Loading Dose + 24-hour IV infusion (3.5 mg/hour).

DETAILED DESCRIPTION:
This will be a single center, open-label phase 1 study in healthy Chinese subjects. A total of up to 16 subjects may be enrolled to achieve a total target of 12 evaluable subjects.

Subjects will remain in-house for the entire study. All subjects will be discharged at End-of-Study (EOS) on Day 5.

A full dose for NTM-001 will be defined as a 12.5 mg IV Loading Dose + 24-hour IV infusion (3.5 mg/hour).

Subjects who withdraw or are withdrawn from the study will not be replaced since attrition is considered.

Blood will be collected for PK analysis. Safety assessments will include the following: adverse events (AEs), vital sign measurements, physical examinations, 12-lead electrocardiograms (ECGs), and clinical laboratory evaluations. infusion site reactions will be recorded as AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female Chinese with his/her biological parents and grandparents are of Chinese ethnicity, aged 18 to 45 years, inclusive at Screening.
2. Subject has a body mass index (BMI) between 19.0 and 24.0 kg/m2 at Screening and Baseline.
3. Subject has a body weight ≥50 kg at Screening and Baseline.
4. Subject is in good health, as determined by the Investigator, based on medical history, no findings of clinical significant abnormalities at physical examination, vital signs and clinical laboratory tests at Screening and Baseline.
5. Subject has normal renal function (CrCl ≥ 90 mL/min) as determined by Cockcroft Gault formula at Screening and Baseline.
6. Negative blood pregnancy test at Screening and negative urine test at Baseline for women of childbearing potential (WOCBP). For the purposes of this study, WOCBP is defined as: "All female subjects after puberty unless they are postmenopausal for at least 24 months, are surgically sterile for at least 6 months, or are sexually inactive for at least 6 weeks prior to first dose and throughout the study".
7. Subject is able to communicate well with the Investigator and is willing to comply with the requirements of the entire study.
8. Subject provides a written informed consent prior to the performance of any study procedure.

Exclusion Criteria:

1. Subject has known hypersensitivity to ketorolac or any of the excipients in the Test or Reference formulations
2. There is evidence in the subject's medical history or in the medical examination or clinical laboratory results of any clinically significant hepatic, renal, gastrointestinal, cardiovascular, pulmonary, hematological or other significant acute or chronic abnormalities which might influence either the safety of the subject, interfere with trial procedures or outcomes, explicitly the absorption, distribution, metabolism or excretion of the active agent under investigation.
3. Subjects who smoked more than 5 cigarettes per day during the 3 months prior to screening or did not agree to refrain from using any tobacco products during the study period.
4. Subject has significant acute or chronic infections, including, among others:

   1. Known history of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome or HIV antibody positive.
   2. Hepatitis B virus (HBV) surface antigen positive or Hepatitis C virus (HCV) antibody positive.
   3. Active tuberculosis (history of exposure or history of positive tuberculin test, plus, presence of clinical symptoms, physical or radiographic findings). If the Investigator suspects a potential risk history for tuberculosis, the physician may use the Quanteferon® test to omit the risk.
5. Subject has chronic malnutrition or severe hypovolemia.
6. Subject is pregnant or breastfeeding. Pregnancy status will be confirmed by serum assay for qualitative human chorionic gonadotropin (hCG) at Screening and urine assay at Baseline for females of child-bearing potential.
7. Subject has a positive test result for amphetamines including methylenedioxymethamphetamine and methamphetamine, barbiturates, benzodiazepines, cocaine, marijuana (THC), opioids including opiates and methadone or alcohol (blood) at Screening or Baseline.
8. Subject has a history of any drug or alcohol abuse in the past 2 years or alcohol consumption greater than 21 units per week. A unit of alcohol will be equivalent to 1 can of beer, 1 glass of wine, or the equivalent of 1 alcoholic drink. Alcohol consumption is prohibited within 96 hours before entry to the study site on Day -1 and throughout the entire study until discharge.
9. Subject has donated or lost greater than 50 mL of blood in the 3 months prior to the administration of the first dose of study drug.
10. Subject has taken or will need taking any prescription or nonprescription drugs (including vitamins and dietary or herbal supplements) within 2 weeks before the start of study treatment until completion of the end of study/early termination visit or 5 half-lives of investigational drug, whichever was longer.
11. Subject has been administered a live vaccine within 28 days prior to study entry.
12. Subject has contacted with a confirmed or suspected COVID-19 patient within 14 days prior to screening.
13. Subject has current or past clinical study participation in the past 3 months or within 5 half-lives of the investigational drug, whichever was greater.
14. Subject has any medical condition wherein the Investigator determines the subject is not suited for this study, including but not limited to subjects who have conditions that are contraindicated as outlined in the ketorolac product label such as:

    1. A history of peptic ulcer disease or gastrointestinal bleeding or perforation oractive peptic ulcer disease
    2. A history of asthma, urticaria or allergic-type reactions after taking aspirin or other NSAIDs
    3. History of, or suspected or confirmed cerebrovascular bleeding, hemorrhagic diathesis, incomplete hemostasis
    4. Increased risk of bleeding at the discretion of the investigator based on prior/concomitant disease, laboratory values, use of the medication with anticoagulation effect (such as warfarin) or surgical complication
    5. Risk for renal failure due to volume depletion
    6. Concomitant use of aspirin or NSAID, probenecid or pentoxifylline
15. Subject is institutionalized.
16. Subject has any psychiatric condition that would prohibit the understanding or rendering of informed consent or that would limit compliance with study requirements.
17. Females of childbearing potential refuse to use one of the following acceptable birth control methods:

    1. IUD in place for at least 3 months prior to entering the study;
    2. barrier methods (as condom or diaphragm) with spermicide for at least 28 days prior to the first dose and throughout the study;
    3. surgical sterilization of the partner (vasectomy for 6 months minimum prior to the patient's entering the study);
    4. hormonal contraception for at least 3 months prior to the first dose of study drug. Postmenopausal women must have reported amenorrhea for at least 2 years.
18. Male subjects who are apt to procreate refuse to use an acceptable contraceptive regimen during the entire study, and until at least 90 days after the drug administration.
19. Study site personnel or sponsor's employees are NOT allowed to participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Cmax of NTM-001 | 0 to 96 hours
  Maximum observed plasma concentration (Cmax).
AUC0-t of NTM-001 | 0 to 96 hours
  Area under the plasma concentration-versus-time curve from time 0 to the last collection time after drug administration with a concentration equal to or greater than the lower limit of quantification (AUC0-t).
AUC0-∞ of NTM-001 | 0 to 96 hours
  Area under the plasma concentration-versus-time curve from time 0 extrapolated to infinity after drug administration (AUC0-∞).
Tmax of NTM-001 | 0 to 96 hours
  Time to maximum observed plasma concentration (Tmax).
t1/2 of NTM-001 | 0 to 96 hours
  Apparent terminal elimination half-life (t1/2).

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Cheung, Doctor, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- HUK Phase 1 clinical trials center, Hong Kong, Hong Kong, China